CLINICAL TRIAL: NCT00482716
Title: Randomized Controlled Study of Iron Supplementation to Support the Response to Recombinant Human Erythropoietin for the Treatment of Chemotherapy-Induced Anaemia
Brief Title: Epoetin Alfa or Epoetin Beta With or Without Iron Infusion in Treating Anemia in Patients With Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Bartholomew's Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000549549; BARTS-06/Q0605/93; ISRCTN11830961; EU-20731
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2009-08

CONDITIONS: Anemia; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage I marginal zone lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; anemia
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Epoetin Alfa; epoetin beta; Iron-Dextran Complex; Ferric Oxide, Saccharated

INTERVENTIONS:
Biological: epoetin alfa
Biological: epoetin beta
Dietary Supplement: iron dextran complex
Dietary Supplement: iron sucrose injection

SUMMARY:
RATIONALE: Epoetin alfa and epoetin beta may cause the body to make more red blood cells. Red blood cells contain iron that is needed to carry oxygen to the tissues. It is not yet known whether epoetin alfa or epoetin beta are more effective when given with or without iron infusion in treating anemia in patients with cancer.

PURPOSE: This randomized phase III trial is studying epoetin alfa or epoetin beta to compare how well they work with or without iron infusion in treating anemia in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of recombinant epoetin alfa or epoetin beta with vs without parenteral iron in anemic, iron-replete patients with nonmyeloid malignancies.

OUTLINE: This is a randomized, controlled, open-label, prospective study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive recombinant erythropoietic stimulatory activity (ESA) therapy comprising epoetin alfa or epoetin beta subcutaneously (SC) on day 1.
* Arm II: Patients receive ESA therapy as in arm I and parenteral iron (i.e., low molecular weight iron dextran complex IV over 5-10 minutes or iron sucrose injection IV over 10-30 minutes) on day 1.

In both arms, treatment repeats weekly for up to 10 weeks or until hemoglobin reaches 13 g/dL, whichever comes first.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of nonmyeloid malignancy

  * No primary bone marrow malignancies except multiple myeloma, chronic lymphocytic leukemia, or indolent non-Hodgkin lymphoma
* Candidate for erythropoietin stimulatory activity therapy for anemia due to cancer and/or chemotherapy

  * Baseline hemoglobin ≤ 10.5 g/dL
  * Planning to receive ≥ 6 additional weeks of chemotherapy for the malignancy
* Demonstrates iron-replete status as defined by all of the following parameters:

  * Percent saturation of transferrin ≥ 20%
  * Serum ferritin 225-2,250 pmol/L
  * Reticulocyte hemoglobin content > 31 pg
  * Zinc protoporphyrin < 80 µg/dL
* No anemia of origin other than cancer or cancer chemotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* No allergy or intolerance to recombinant epoetin alfa or epoetin beta
* No known sensitivity to iron sucrose injection or iron dextran complex
* No uncontrolled hypertension
* No active infection
* No active bleeding

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior iron sucrose injection or iron dextran complex therapy
* More than 6 months since prior and no concurrent transfusion

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-01

PRIMARY OUTCOMES:
Maximum hemoglobin achieved

SECONDARY OUTCOMES:
Time to zenith hemoglobin or achievement of hemoglobin level ≥ 13 g/dL

CONTACTS AND LOCATIONS:
Overall Officials: Samir G Agrawal, MD, PhD, Study Chair — St. Bartholomew's Hospital
Locations (1):
- Saint Bartholomew's Hospital, London, England, United Kingdom